CLINICAL TRIAL: NCT02306954
Title: Phase II Randomized Study of High Dose Interleukin-2 Versus Stereotactic Body Radiation (SBRT) and High Dose Interleukin-2 (IL-2) in Patients With Metastatic Renal Cancer
Brief Title: Study of High Dose Interleukin-2 (IL-2) and Stereotactic Body Radiation (SBRT) in Patients With Metastatic Renal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: Prometheus Laboratories (Industry); Cytokine Working Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 14-256A
Record Dates: First submitted 2014-11-30; First posted 2014-12-03 (Estimated); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Renal Cell Carcinoma
Keywords: Kidney Cancer; High Dose IL-2; SBRT
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Dose IL-2 (Active Comparator): Patients will receive IL-2 at 600,000 international units per kg IVB every 8 hours for 14 planned doses with an additional cycle 14 days after the first. Responding patients with regressing disease are eligible for up to 6 IL-2 cycles.
  Patients assigned to the IL-2 arm who have disease progression after the first two IL-2 cycles have the option to receive SBRT followed by 2 additional cycles of IL-2.
  Interventions: Biological: High Dose IL-2
- High Dose IL-2 and SBRT (Experimental): Patients assigned to SBRT arm will receive two doses of SBRT at 20 Gy on the Wednesday and Friday before IL-2 starts (the following Monday). Patients will receive IL-2 at 600,000 international units per kg IVB every 8 hours for14 planned doses with an additional cycle 14 days after the first. Responding patients with regressing disease are eligible for up to 6 IL-2 cycles.
  Interventions: Biological: High Dose IL-2; Radiation: SBRT

INTERVENTIONS:
Biological: High Dose IL-2 — High Dose IL-2 is approved by the FDA for the treatment of renal cell cancer.
  Other Names: Proleukin
Radiation: SBRT — Patients assigned to SBRT arm will receive two doses of SBRT at 20 Gy on the Wednesday and Friday before the Monday on which IL-2 starts.
  Arms: High Dose IL-2 and SBRT

SUMMARY:
All patients will receive IL-2 (14 planned doses with an additional cycle 14 days after the first). Responding patients with regressing disease are eligible for up to 6 IL-2 cycles. Patients assigned to SBRT arm will receive two doses of SBRT on the Wednesday and Friday before the Monday on which IL-2 starts.

DETAILED DESCRIPTION:
All patients will receive IL-2 at 600,000 international units per kilogram (kg) by intraveneous bolus (IVB) every 8 hours for 14 planned doses with an additional cycle 14 days after the first. Responding patients with regressing disease are eligible for up to 6 IL-2 cycles. Patients assigned to SBRT arm will receive two doses of SBRT at 20 Gray (Gy) on the Wednesday and Friday before the Monday on which IL-2 starts.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of predominant conventional (clear cell) renal cancer
* Patients must be ≥ 18 years of age
* Tumors amenable to SBRT in lungs (central locations preferred), mediastinum, chest wall, bones with a soft tissue component (other than long bones), or liver, liver hilum and associated lymph nodes (inclusive of immediately adjacent masses), 1 - 3 foci; no minimum size, but none greater than 7 cm. Patients may have other metastases but only a maximum of 3 will be treated
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Women of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to the start of protocol treatment. In addition, women of childbearing potential as well as male patients must agree to take appropriate precautions to avoid pregnancy
* Patients must agree to participate in the Prometheus IL-2 patient registry (PROCLAIM registry)
* Patients must sign a study-specific consent form

Exclusion Criteria:

* No metastatic site amenable to SBRT
* Patients with brain metastases not candidates for radiosurgery alone
* Previous radiation to sites proposed for SBRT
* Patients with active systemic, pulmonary, or pericardial infection
* Pregnant or lactating women, as treatment involves unforeseeable risks to the embryo or fetus
* Evidence of ischemia on exercise tolerance test, stress thallium study, or baseline EKG
* Clinically significant underlying pulmonary disease as measured by pulmonary function tests
* Blood tests within protocol-specified range
* Need for chronic steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2014-12; Primary Completion 2020-09-15 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Response Rate | 5 years
  The objective of this study is to compare the response rate among renal cell cancer (RCC) patients of high dose IL-2 to SBRT + IL-2 in patients with metastatic renal cancer

SECONDARY OUTCOMES:
Response Rate in Patients Who Receive SBRT following Progression on IL-2 | 5 years
  Measure the response of SBRT + IL-2 in patients with RCC who have disease progression after high-dose IL-2

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Curti, MD, Principal Investigator — Providence Health & Services
Locations (1):
- Portland Providence Medical Center, Portland, Oregon, United States

REFERENCES:
- See also: Providence Cancer Center — http://oregon.providence.org/our-services/p/providence-cancer-center/